CLINICAL TRIAL: NCT06713668
Title: Augmented Pacing for Shock in the Cardiac Intensive Care Unit - A Pilot Patient-level Crossover Trial
Brief Title: Augmented Pacing for Shock in the Cardiac Intensive Care Unit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, JGarry, Cardiovascular Medicine Research Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 241410
Record Dates: First submitted 2024-11-01; First posted 2024-12-03 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Cardiogenic Shock; Bradycardia; Shock
Keywords: Cardiogenic Shock; Bradycardia; Shock; Pacing
MeSH Terms: conditions — Shock, Cardiogenic; Bradycardia; Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Pacing (75 bpm) then Augmented Pacing (100 bpm) (Other): Backup pacing rate will be set to 75 bpm first then 100 bpm second
  Interventions: Device: Backup Pacing Rate Change
- Augmented Pacing Rate (100 bpm) then Standard Pacing (75 bpm) (Other): Backup pacing rate will be set to 100 bpm first then 75 bpm second
  Interventions: Device: Backup Pacing Rate Change

INTERVENTIONS:
Device: Backup Pacing Rate Change — Patients will have backup pacing programmed to A (75 bpm) and B (100 bpm), randomizing to sequence of exposure A-B or B-A

SUMMARY:
The goal of this clinical trial is to learn if backup pacing at an increased rate improves hemodynamics in adults with relative bradycardia, a permanent pacemaker, and cardiogenic shock. The main question it aims to answer is:

Does increasing the backup pacing rate to 100 beats per minute lead to improved cardiac index compared to a backup pacing rate of 75 beats per minute

Participants who are already hospitalized in the Cardiovascular Intensive Care Unit with a permanent pacemaker and pulmonary artery catheter in place will be enrolled in this study. Participants will be exposed to each pacemaker rate in a randomized order with hemodynamics assessed after 10 minutes at each rate.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 and older)
* Located in the CVICU
* FDA approved permanent pacemaker in place (inclusive of dual-chamber and Bi-Ventricular ICDs) with labeling that allows backup pacing setting at 100 bpm.
* Receiving a vasopressor or Inotrope for at least 4 hours
* Average HR ≤ 75 bpm over the last hour (on Telemetry review)
* Pulmonary artery catheter in place with functioning thermistor and pulmonary artery port.

Exclusion Criteria:

* Single chamber Implantable Cardiac Defibrillator
* Sinus rhythm with a leadless pacemaker
* Ventricular Tachycardia or Ventricular Fibrillation arrest in last 48 hours
* Hemodynamic instability within the last 4 hours, defined as an increase in the dose of norepinephrine > 10 mcg/min, an increase of epinephrine > 10 mcg/kg/min, or initiation of a second vasopressor
* Alternative indication for pacing rate change (i.e Torsade de Pointes, Recurrent Ventricular Tachycardia)
* Comfort-focused care or anticipated death within 24 hours
* Mechanical circulatory support in place
* Newly discovered pacing system malfunction (lead displacement, loss of capture, elevated capture threshold, significant lead impedance change, battery depletion, undersensing or oversensing)
* Non-English Speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-04-22 (Estimated); Study Completion 2027-04-22 (Estimated)

PRIMARY OUTCOMES:
Cardiac Index by thermodilution | At baseline and 10 minutes after each rate programmed (i.e at 0, 15, and 30 minutes)
  Cardiac Index measured by thermodilution (in liters per minute per meters squared)

SECONDARY OUTCOMES:
Cardiac Index by Indirect Fick | 0, 15, 30 minutes.
Cardiac Output by thermodilution | 0, 15, 30 minutes.
Cardiac Output by indirect fick | 0 ,15, 30 minutes
Central Venous Pressure | 0, 15, 30 minutes
Pulmonary Artery Systolic Pressure | 0, 15, 30 minutes
Pulmonary Artery Diastolic Pressure | 0, 15, 30 minutes
Pulmonary Artery Pulsitility Index | 0, 15, 30 minutes
Right Ventricular Stroke Work Index | 0, 15, 30 minutes
Pulmonary Artery (Mixed Venous) Blood Hemoglobin saturation | 0, 15, 30 minutes
Cardiac Power Index (Thermodilution and indirect fick) | 0, 15, 30 minutes
Cardiac Power Output (Thermodilution and indirect fick) | 0, 15, 30 minutes
Systolic Blood pressure | 0, 15, 30 minutes
Diastolic Blood Pressure | 0, 15, 30 minutes
Mean Arterial Pressure | 0, 15, 30 minutes
Difference in vasopressor/inotrope requirements | 0, 15, 30 minutes
Arrhythmia events (Atrial and Ventricular) | 0, 15, 30 minutes
Percentage of PVCs | 0, 15, 30 minutes
Pacing percentage (Atrial, RV or Bi-V) | 0, 15, 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No